CLINICAL TRIAL: NCT00929903
Title: A Phase I Study of Pazopanib as a Single Agent for Children With Relapsed or Refractory Solid Tumors
Brief Title: Pazopanib Hydrochloride in Treating Young Patients With Solid Tumors That Have Relapsed or Not Responded to Treatment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01929; NCI-2011-01929 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ADVL0815; CDR0000646720; ADVL0815 (Other: COG Phase I Consortium); ADVL0815 (Other: CTEP); U01CA097452 (NIH)
Record Dates: First submitted 2009-06-27; First posted 2009-06-30 (Estimated); Last update posted 2013-09-30 (Estimated); Status verified 2013-09

CONDITIONS: Childhood Central Nervous System Choriocarcinoma; Childhood Central Nervous System Embryonal Tumor; Childhood Central Nervous System Germ Cell Tumor; Childhood Central Nervous System Germinoma; Childhood Central Nervous System Mixed Germ Cell Tumor; Childhood Central Nervous System Teratoma; Childhood Central Nervous System Yolk Sac Tumor; Metastatic Childhood Soft Tissue Sarcoma; Recurrent Childhood Brain Stem Glioma; Recurrent Childhood Central Nervous System Embryonal Tumor; Recurrent Childhood Soft Tissue Sarcoma; Recurrent Childhood Visual Pathway Glioma; Unspecified Childhood Solid Tumor, Protocol Specific
MeSH Terms: conditions — Optic Nerve Glioma | interventions — pazopanib

ARMS (1):
- Treatment (pazopanib hydrochloride) (Experimental): Patients receive oral pazopanib hydrochloride once daily on days 1-28. Courses repeat every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: pazopanib hydrochloride; Other: pharmacological study

INTERVENTIONS:
Drug: pazopanib hydrochloride — Given orally
  Other Names: GW786034B; Votrient
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of pazopanib hydrochloride in treating young patients with solid tumors that have relapsed or not responded to treatment. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the maximum-tolerated dose and/or recommended phase II dose of pazopanib hydrochloride in pediatric patients with relapsed or refractory solid tumors.

II. Define and describe the toxicities of this regimen in these patients. III. Characterize the pharmacokinetics of pazopanib hydrochloride in these patients.

SECONDARY OBJECTIVES:

I. Preliminarily define the antitumor activity of pazopanib hydrochloride within the confines of a phase I study.

II. Evaluate changes in tumor vascular permeability following initiation of pazopanib hydrochloride and correlate these changes with clinical outcome by dynamic contrast-enhanced MRI.

OUTLINE: This is a multicenter study dose-escalation study.

Patients receive oral pazopanib hydrochloride once daily on days 1-28. Courses repeat every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity. Patients accrued after the maximum-tolerated dose (MTD) of pazopanib hydrochloride has been determined receive pazopanib hydrochloride as an oral suspension.

Some patients undergo dynamic contrast-enhanced MRI at baseline and periodically during study. Blood samples are collected at baseline and periodically during study for pharmacokinetic studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

NOTE: Histologic confirmation not required for intrinsic brain stem cell tumor, optic pathway gliomas, pineal tumors and elevations of cerebrospinal fluid, and serum tumor markers including alpha-fetoprotein or beta-human chorionic gonadotropin.

* Histologically confirmed relapsed or refractory solid tumors at original diagnosis including CNS tumors* (Part 1 and Part 2a)

  * Neurologic deficits in patients with CNS tumors must have been relatively stable for ≥ 1 week
* Histologically confirmed soft tissue sarcoma, desmoplastic small round cell tumor, or extraosseus Ewing sarcoma at original diagnosis including the following (Part 2b):

  * Tumor in the head, neck, or extremity or fixed within the abdomen or pelvis that it is not sensitive to motion artifact
  * No isolated pulmonary metastases

    * Disease with no known curative therapy or no therapy proven to prolong survival with acceptable quality of life
    * Measurable or evaluable disease (Part 1 and Part 2a)
    * Measurable tumor that is ≥ 2 cm in its longest diameter (Part 2b)
    * Patients must be:
* > 2 years of age and ≤ 21 years of age (Part 1 and Part 2a)
* > 2 years of age and ≤ 25 years of age (Part 2b)

  * Body surface area ≥ 0.48 m^2 (Part 1 and Part 2b)
  * For patients with CNS tumors or CNS metastasis, there must be no evidence of new CNS hemorrhage of more than punctate size and/or > 3 foci of punctate hemorrhage on baseline MRI for primary CNS tumors ≥ 14 days prior to study entry
  * Karnofsky performance status (PS) 50-100% (> 16 years of age)
  * Lansky PS 50-100% (≤ 16 years of age)
  * Platelet count ≥ 100,000/mm^3 (transfusion independent)
  * ANC ≥ 1,000/mm^3
  * Hemoglobin ≥ 8.0 g/dL (may receive RBC transfusions)
  * Creatinine clearance or radioisotope GFR ≥ 70 mL/min OR serum creatinine based on age/gender as follows:
* 0.6 mg/dL (1 to < 2 years of age)
* 0.8 mg/dL (2 to < 6 years of age)
* 1 mg/dL (6 to < 10 years of age)
* 1.2 mg/dL (10 to < 13 years of age)
* 1.5 mg/dL (male ) or 1.4 mg/dL (female) (13 to < 16 years of age)
* 1.7 mg/dL (male) or 1.4 mg/dL (female) ( ≥ 16 years of age)

  * Urine protein:creatinine ratio < 1 OR urinalysis negative for protein OR 24-hour urine protein level < 1 g
  * Bilirubin ≤ 1.5 times upper limit of normal (ULN)
  * ALT ≤ 110 U/L
  * PT and PTT ≤ 1.2 times ULN
  * INR ≤ 1.2
  * Serum albumin ≥ 2 g/dL
  * No grade > 1 abnormalities of potassium, calcium, magnesium, or phosphorous
* Supplementation allowed

  * Not pregnant or nursing
  * Negative pregnancy test
  * Fertile patients must use effective contraception
* Oral contraceptives are not considered effective

  * Adequate cardiac function defined as any of the following:
* Shortening fraction of ≥ 27% by echocardiogram
* Ejection fraction of ≥ 50% by gated radionuclide study
* QTc < 450 msec
* No history of myocardial infarction, severe or unstable angina, or peripheral vascular disease or familial QTc prolongation

  * Adequate blood pressure defined as ≤ 95th percentile for age, height, and gender
  * Known history of well-controlled seizures allowed
  * Able to swallow whole tablets (Part 1 and Part 2b)
  * No uncontrolled infection
  * No evidence of active bleeding, intratumoral hemorrhage, or bleeding diathesis
  * None of the following conditions within the past 6 months:
* Arterial thromboembolic events, including transient ischemic attack or cerebrovascular accident
* Pulmonary embolism
* Deep vein thrombosis
* Other venous thromboembolic event

  * No hemoptysis within the past 6 weeks
  * No serious or non-healing wound, ulcer, or bone fracture
  * No significant traumatic injury within the past 28 days
  * No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
  * No patients who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study
  * No fine-needle aspiration within 48 hours before day 1 of therapy
  * Fully recovered from all prior therapy (e.g., chemotherapy, immunotherapy, or radiotherapy)
  * At least 3 weeks since prior myelosuppressive chemotherapy (6 weeks for prior nitrosourea)
  * At least 7 days since prior hematopoietic growth factor
  * At least 21 days since prior VEGF-Trap
  * No prior pazopanib hydrochloride
  * At least 7 days since prior VEGF-blocking tyrosine kinase inhibitor or other biological agents
  * At least 3 half-lives since prior monoclonal antibody, including bevacizumab
  * At least 21 days since any other prior anticancer antibody therapy
  * At least 2 weeks since prior local palliative radiotherapy (small port)
  * At least 3 months since prior total-body irradiation, craniospinal radiotherapy, or ≥ 50% radiotherapy to the pelvis
  * At least 6 weeks since prior other substantial bone marrow radiotherapy
  * At least 2 months since stem cell transplantation and no evidence of graft-vs-host disease
  * Thyroid replacement therapy allowed provided a stable dose has been received for ≥ 4 weeks
  * No concurrent medication for cardiac function or hypertension
  * Concurrent corticosteroids allowed provided dose is stable or decreasing for > 7 days (for patients enrolled in Part 1 and Part 2a of study)
* No concurrent corticosteroids for patients enrolled in Part 2b of the study

  * No other concurrent anticancer agents or radiotherapy
  * No other concurrent investigational drugs
  * No concurrent enzyme-inducing anticonvulsants
  * No concurrent anticoagulation therapy with coumadin and/or low molecular weight heparin
* Prophylactic anticoagulation therapy (i.e., intraluminal heparin) of venous or arterial access devices allowed

  * No concurrent aspirin, ibuprofen, or other NSAIDs
  * No concurrent drugs metabolized through several of the specific P450 cytochrome isoform including inducers or inhibitors of CYP3A4
  * No concurrent drugs with a known risk of torsades de pointes
  * At least 28 days since prior major surgical procedure, laparoscopic procedure, or open biopsy
* Port placement or central line placement 48 hours before day 1 of therapy allowed

  * No core biopsy within the past 7 days

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2009-06; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose of pazopanib hydrochloride defined as the maximum dose at which fewer that one-third of patients experience DLT | 28 days
  Graded using the NCI CTCAE version 4.0.
Adverse events according to NCI CTCAE version 4.0 | Up to 30 days after completion of study treatment
Pharmacokinetics of pazopanib hydrochloride | Baseline, days 15, 22, and 27 of course 1 and day 1 of odd courses
  Summarized with simple summary statistics, including means, medians, ranges, and standard deviations (if numbers and distribution permit).

SECONDARY OUTCOMES:
Overall response to pazopanib hydrochloride according to RECIST criteria | Up to 30 days after completion of study treatment
  The overall response assessment takes into account response in both target and non-target lesions, the appearance of new lesions and normalization of markers.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Glade-Bender, Principal Investigator — COG Phase I Consortium
Locations (14):
- United States (14):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Indiana University Medical Center, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

REFERENCES:
- [Derived] Glade Bender JL, Lee A, Reid JM, Baruchel S, Roberts T, Voss SD, Wu B, Ahern CH, Ingle AM, Harris P, Weigel BJ, Blaney SM. Phase I pharmacokinetic and pharmacodynamic study of pazopanib in children with soft tissue sarcoma and other refractory solid tumors: a children's oncology group phase I consortium report. J Clin Oncol. 2013 Aug 20;31(24):3034-43. doi: 10.1200/JCO.2012.47.0914. Epub 2013 Jul 15. PMID 23857966